CLINICAL TRIAL: NCT00690014
Title: Evaluation of Renal Drug Transport in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-26129; 1R15GM072526-01 (NIH)
Record Dates: First submitted 2008-06-02; First posted 2008-06-04 (Estimated); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Kidney Disease
Keywords: OAT; GFR; renal function; PAH
MeSH Terms: conditions — Kidney Diseases | interventions — Probenecid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental)
  Interventions: Drug: probenecid

INTERVENTIONS:
Drug: probenecid — 500 mg q 6 hrs

SUMMARY:
The process of drug elimination that occurs within the kidneys is complex, and involves filtration, secretion and absorptive mechanisms. Many drugs, metabolites and toxins, including organic anions and cations, rely on renal mechanisms for elimination from the body. Failure to recognize the contribution of renal mechanisms involved in drug elimination during the drug development process can result in drug interactions or toxicity in clinical trials. This is increasingly important due to the use of OAT1 inhibitors such as probenecid that are being used in adjuvant treatment regimens. Thus, in order to more fully understand the effects renal disease, drugs and nephrotoxins on the renal transport pathways of tubular secretion in humans, novel approaches that incorporate both in vitro (experimental) as well as clinical observations (clinical trial), also called in-vitro/in-vivo correlations (IVIVC) need to be developed. These methods can then be used to identify and evaluate specific kidney "probe" drugs that undergo extensive tubular secretion. Such approaches are needed to characterize drug clearance by tubular mechanisms and to identify potentially significant drug-drug interactions prior to exposure to patients in Phase 2 and 3 clinical trials. This investigator-initiated pilot project aims to determine the pharmacokinetics of selected FDA-approved compounds (PAH, iothalamate) for use in IVIVC model development. The proposed research is innovative, because it involves a translational approach to development of an IVIVC model applied to renal drug clearance. It is our expectation that the resultant approach will further our understanding of pharmacogenomics, inter-subject variability and renal drug clearance. This approach will generate important new information regarding in vitro drug-drug interactions in light of many new and potent OAT1 blocking agents being introduced for the treatment of human diseases. In future studies, we hope to fully characterize the effects of diseases such as diabetes, hypertension, and nephropathy on renal drug transport mechanisms using IVIVC models. We expect that results from this NIH-funded study will provide needed preliminary data to design future pharmacogenomic and drug interaction studies in humans.

DETAILED DESCRIPTION:
The purpose of this study is to measure GFR (using iothalamate clearance) and renal tubular function (using PAH clearance) in healthy subjects. The protocol will be approved by the University of Maryland IRB and the General Clinical Research Center (GCRC) advisory committee (GAC). Following the informed consent process, each subject will be evaluated for past medical history, undergo a physical examination and routine laboratory tests (including urinary protein:creatinine ratio) conducted within 1 month prior to the study visit.

Day 1: Vital signs (heart rate, blood pressure, respiratory rate) will be recorded hourly throughout each study visit. Subjects will have intravenous catheters inserted into forearm veins of each arm for blood collection and intravenous infusion iothalamate and PAH. From 30 minutes before marker administration until the end of each evaluation period, subjects will remain in a semireclined position except during urine collections. A constant-rate infusion will then be initiated at 1 mL/min for a total of 3 hours, with the concentration in the infusate determined based on the patient's estimated renal clearance and target plasma concentration of 10 mg/L and 15 mg/L for iothalamate, and PAH, respectively. Day 2: Washout Day 3: Subject will begin taking probenecid. Day 4 (Study visit #2): Subject will be admitted to the GCRC at 8AM. The final dose of probenecid will be administered. The renal function test will then be conducted as described for study visit #1 above. Day 11: Subject will be contacted for monitoring of adverse events according to GCRC procedures.

ELIGIBILITY:
Inclusion Criteria:

* Adult, aged 18 to 40 years
* Healthy based on review of past medical history and physical examination (normal biochemical screen and urinalysis)
* Signed inform consent

Exclusion Criteria:

* Any medications taken within 48 hours prior to study
* History of gout or gouty arthritis
* History of uric acid
* Kidney stones
* History of known allergic or adverse reactions to diagnostic iodine containing compounds including iothalamate, PAH or probenecid, will be excluded.
* Subjects with current or preexisting liver disease (including hepatitis) as evidenced by elevated INR, liver transaminases (AST/ALT), bilirubin, or serum albumin < 3.0 g/dL.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2006-08 (Actual); Primary Completion 2007-04 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Effect of probenecid on renal clearance of PAH (renal function probe) | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Dowling, PhD, Principal Investigator — University of Maryland, College Park
Locations (1):
- University of Maryland GCRC, Baltimore, Maryland, United States